CLINICAL TRIAL: NCT01180153
Title: An Pilot Study of S-1 Combined With Oxaliplatin for First-line Treatment of Unresectable, Metastatic or Locally Advanced Biliary Tract Cancer or Ampullary Adenocarcinoma
Brief Title: Study of S-1 Oxaliplatin (SOX) for Biliary Tract Cancer (BTC) (Ampullary Adenocarcinoma)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Lin Shen, Beijing Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChinaBJCH_SOX_BTC
Record Dates: First submitted 2010-08-09; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Biliary Tract Cancer
Keywords: 40 S-1/L-OHP; biliary tract; ampullary carcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOX: advanced BTC or ampullary carcinoma (Experimental): unresectable, metastatic or locally advanced biliary tract or ampullary adenocarcinoma receive SOX regimen
  Interventions: Drug: S-1 oxaliplatin

INTERVENTIONS:
Drug: S-1 oxaliplatin — S-1 (20mg, 25mg); L-OHP (50 mg)
  Other Names: S-1 (20mg, 25mg); L-OHP (50 mg)

SUMMARY:
To evaluate efficacy and safety of S-1 Oxaliplatin (SOX) regimen to patients with unresectable, metastatic or locally advanced biliary tract or ampullary adenocarcinoma.

DETAILED DESCRIPTION:
To list in cases with unresectable, metastatic or locally advanced biliary tract or ampullary adenocarcinoma that have not been treated before,confirm the efficacy and safety of combined S-1/L-OHP regimen for the biliary tract or ampullary carcinoma, providing evidence-based proof for the future treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed by the subject itself;
2. Aged over 18;
3. With a definite pathological or cytological diagnosis of adenocarcinoma;
4. No pre-treatment (including radiotherapy, chemotherapy, immunotherapy, etc.). For recurrent cases, if the subjects have received adjuvant chemotherapy without S-1 or L-OHP after surgery and the time to the end date of adjuvant chemotherapy is over 6 months, they can also be enrolled;
5. Enhanced helical CT or MRI scanning shows a target lesion over 1cm within 14 days before enrollment
6. Within 7 days before enrollment, baseline blood routine and biochemical indicators meet the following criteria:

   * Hemoglobin ≥ 90g/L,
   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L,
   * Platelets ≥ 100×109/L，
   * Serum total bilirubin < 1.5 times of the upper normal limit,
   * Serum creatinine < upper limit of normal,
   * Serum albumin ≥ 30 g/L;
7. Can receive oral administration;
8. Karnofsky(KPS) score ≥ 70 points;
9. Expected survival time is more than 90 days;
10. Women of childbearing age must receive urine or blood pregnancy test within 7 days before randomization and the results are negative;
11. Male and female patients of appropriate reproductive age are willing to use reliable contraception methods for contraception in the process of study till 30 days after drug withdrawal.

Exclusion Criteria:

1. Patients with a severe drug allergy history (including mildly allergic to L-OHP, 5-FU, FT207, 5-HT3 receptor antagonist);
2. Patients who participated or are participating in other clinical trials within 4 weeks before enrollment;
3. Patients who have received blood transfusion, blood products and hematopoietic factor preparations such as G-CSF within 15 days before enrollment;
4. Patients who have undergone a surgery within 15 days before enrollment, and its effects have not been eliminated;
5. Patients with diarrhea;
6. Patients with a complication of active infection (infection causes a fever above 38 ℃);
7. Patients accompanied by dysphagia, complete or incomplete gastrointestinal obstruction, active gastrointestinal bleeding and perforation, etc. that cause difficulty in taking S-1 orally;
8. Patients with severe liver disease (e.g. active hepatitis, cirrhosis, etc.), renal insufficiency, severe lung disease (interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc.), or uncontrollable diabetes, hypertension and other chronic systemic diseases;
9. Patients who have received long-term systemic steroid therapy (Note: short-term users with steroid withdrawal > 2 weeks can be selected);
10. Patients with brain metastases or suspected of brain metastases;
11. Patients with peripheral nervous system disorder or a history of significant mental disorder and central nervous system disorder;
12. Heart disease of significant clinical symptoms, e.g. congestive heart failure, coronary heart disease with significant symptoms, arrhythmia and hypertension that are difficult to be controlled by drugs, or with an episode of myocardial infarction within 6 months, or cardiac insufficiency;
13. Patients with pleural effusion, ascites, or pericardial effusion that needs drainage;
14. Pregnant or breast-feeding women, or male and female patients of appropriate reproductive age who refuse to take contraceptive measures;
15. Patients who have suffered from other malignancies within 5 years, except basal cell carcinoma and carcinoma in situ of uterine cervix that have already been cured;
16. Patients without legal capability, or who can not continue the study due to medical or ethical reasons;
17. Patients who are determined not suitable to participate in this clinical trial by the investigators.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 2 years
  to evaluate objective response rate (ORR) of SOX regimen to BTC (Ampullary Adenocarcinoma)

SECONDARY OUTCOMES:
overall survival | 2 years
  to evaluate survival data of overall survival (OS),Progression free Survival(PFS), safety outcome of SOX regimen to BTC (Ampullary Adenocarcinoma)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Professor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Chin Beijing Cancer Hospital, Beijing, Beijing Municipality, China